CLINICAL TRIAL: NCT02406092
Title: An Open-Label, Multinational, Multicenter, Phase IIIB Study to Assess Safety of Rituximab Following Subcutaneous Administration in Patients With CD20+ DLBCL or CD20+ Follicular NHL Grade 1 to 3A
Brief Title: Safety Study of Rituximab (SC) Administered in Participants With CD20+ DLBCL or CD20+ Follicular NHL Grade 1 to 3A
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML28964
Record Dates: First submitted 2015-03-23; First posted 2015-04-02 (Estimated); Results first posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; fludarabine

ARMS (1):
- Rituximab (Experimental): Participants with FL and DLBCL will receive rituximab SC 1400 milligrams (mg) once a month for a minimum of 4 cycles as induction therapy. Participants with FL will continue to receive rituximab once in 2 months for a minimum of 6 cycles as maintenance therapy according to local standards of care. Participants will also receive standard chemotherapy regimen (CHOP [cyclophosphamide+doxorubicin+vincristine+prednisone], CVP [cyclophosphamide+vincristine+prednisone] or FC [fludarabine+cyclophosphamide]) during induction.
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Drug: Fludarabine

INTERVENTIONS:
Drug: Rituximab — Rituximab SC 1400 mg
  Other Names: MabThera®
Drug: Cyclophosphamide — Cyclophosphamide will be administered as per standard local practice.
  Other Names: Endoxan
Drug: Doxorubicin — Doxorubicin will be administered as per standard local practice.
Drug: Vincristine — Vincristine will be administered as per standard local practice.
Drug: Prednisone — Prednisone will be administered as per standard local practice.
Drug: Fludarabine — Fludarabine will be administered as per standard local practice.

SUMMARY:
This open-label, single-arm study will evaluate the safety of rituximab subcutaneously (SC) administered during first line treatment for follicular non-Hodgkin's lymphoma (NHL) (Induction and/or Maintenance treatment plus 24 months of follow up), or diffuse large B-cell lymphoma (DLBCL) (treatment plus 24 months of follow-up).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, cluster of differentiation (CD)20+ DLBCL or CD20+ follicular NHL grade 1 to 3a, according to the world health organization (WHO) classification system
* Currently being treated with rituximab IV in the Induction or Maintenance setting, having received at least one full dose of rituximab IV, defined as standard full dose of rituximab IV 375 milligrams per square meter (mg/m^2) administered without interruption or early discontinuation because of tolerability issues
* Expectation and current ability for the participants to receive at least four additional cycles of treatment during the Induction phase or six additional cycles of treatment during the Maintenance phase (participants with follicular NHL)

Exclusion Criteria:

* Transformed lymphoma or FL IIIB
* History of other malignancy that could affect compliance with the protocol or interpretation of results. This includes a malignancy that has been treated but not with curative intent, unless the malignancy has been in remission without treatment for greater than or equal to (>/=) 5 years prior to dosing

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2015-10-13 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (13):
- Algeria (4):
  - Hôpital Dorban CHU Annaba, Service d'Hématologie, Annaba
  - EHS CAC Hospital FRANTZ FANON ZABANA BLIDA; Hematology ward, Blida
  - EHU Oran, Service d'Hématologie et de Thérapie Cellulaire, Oran
  - Centre hospitalo-univerisitaire de Tizi Ouzou - Nedir Mohamed;Service d'hématologie, Tizi Ouzou
- Morocco (4):
  - CHU 20 Aout Service D'Onco-Hematologie Pediatrique, Casablanca
  - Clinique AlMadina; Service hematologie, Casablanca
  - Centre Hospitalier Uni Ire de Marrakech; Oncologie-Hématologie, Marrakesh
  - Hôpital d'enfants de Rabat - Service d'hémato-oncologie pédiatrique, Rabat
- Tunisia (5):
  - CHU Fattouma Bourguiba, Monastir; Service d'hématologie, Monastir
  - CHU Hédi Chacker; Service d'hématologie, Sfax
  - CHU Farhat Hached; Service d'hématologie, Sousse
  - Aziza Othmana Hospital; Clinical Haematology, Tunis
  - Hopital Militaire d'instruction de Tunis; Service d'hématologie, Tunis

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total of 139 participants mentioned below in the table were recruited and enrolled.
Pre-assignment Details: 139 participants (105 with DLBCL and 34 with FL) in the intent-to-treat (ITT) population; 122 participants (95 with DLBCL and 27 with FL) in the safety population. From 139 participants, 122 were dosed at least 1 dose were included in Safety Analysis Set.
Groups:
- DLBCL Arm: Participants with DLBCL received rituximab SC 1400 milligrams (mg) once a month for a minimum of 4 cycles as induction therapy. Participants with FL will continue to receive rituximab once in 2 months for a minimum of 6 cycles as maintenance therapy according to local standards of care. Participants will also receive standard chemotherapy regimen (CHOP [cyclophosphamide+doxorubicin+vincristine+prednisone], CVP [cyclophosphamide+vincristine+prednisone] or FC [fludarabine+cyclophosphamide]) during induction.
- FL Arm: Participants with FL received rituximab SC 1400 milligrams (mg) once a month for a minimum of 4 cycles as induction therapy. Participants with FL will continue to receive rituximab once in 2 months for a minimum of 6 cycles as maintenance therapy according to local standards of care. Participants will also receive standard chemotherapy regimen (CHOP [cyclophosphamide+doxorubicin+vincristine+prednisone], CVP [cyclophosphamide+vincristine+prednisone] or FC [fludarabine+cyclophosphamide]) during induction.
Period: Overall Study
Arm/Group | DLBCL Arm | FL Arm
Started | 105 | 34
Completed | 67 | 21
Not Completed | 38 | 13
Not completed — Screen failure | 10 | 7
Not completed — Death | 22 | 5
Not completed — Lost to Follow-up | 4 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DLBCL Arm | FL Arm | Total
Number analyzed (Participants) | 105 | 34 | 139
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.3 (13.78) | 52.8 (12.65) | 51.7 (13.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 22 | 78
  Male | 49 | 12 | 61
Race/Ethnicity, Customized [Number; unit: Participants]
  Not Hispanic or Latino | 15 | 4 | 19
  Hispanic or Latino | 0 | 0 | 0
  Other | 74 | 24 | 98
  Not applicable as per local regulations | 16 | 6 | 22

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Administration-Associated Reactions (AARs)
Description: AARs defined as all related adverse events (AEs) occurring within 24 hours of rituximab SC administration, including infusion/injection-related reactions (IIRRs), injection-site reactions, administration site conditions and all symptoms thereof.
Time Frame: Within 24 hours of each rituximab SC administration (maximum treatment duration up to 32 months for FL participants and up to 8 months for DLBCL participants)
Population: Safety Population
Measure: Number; unit: Percentage of Participants %
Groups:
- Overall Population: All participants will receive rituximab SC 1400 milligrams (mg) once a month for a minimum of 4 cycles as induction therapy. Participants with FL will continue to receive rituximab once in 2 months for a minimum of 6 cycles as maintenance therapy according to local standards of care. Participants will also receive standard chemotherapy regimen (CHOP [cyclophosphamide+doxorubicin+vincristine+prednisone], CVP [cyclophosphamide+vincristine+prednisone] or FC [fludarabine+cyclophosphamide]) during induction.
Arm/Group | DLBCL Arm | FL Arm | Overall Population
Number analyzed (Participants) | 95 | 27 | 122
Percentage of Participants %
  Blood And Lymphatic System Disorders, And Lymphatic System Disorders, Anaemia | 1.1 | 3.7 | 1.6
  Blood And Lymphatic System Disorders, Leukopenia | 1.1 | 0 | 0.8
  Blood And Lymphatic System Disorders, Thrombocytopenia | 1.1 | 0 | 0.8
  General Disorders And Administration Site Conditions, Injection Site Erythema | 4.2 | 7.4 | 4.9
  General Disorders And Administration Site Conditions, Injection Site, Injection Site Pain | 4.2 | 0 | 3.3
  Nervous System Disorders, Burning Sensation | 2.1 | 0 | 1.6
  Nervous System Disorders, Paraesthesia | 1.1 | 0 | 0.8
  Skin And Subcutaneous Tissue Disorders, Erythema | 2.1 | 0 | 1.6
  Skin And Subcutaneous Tissue Disorders, Dermatitis Allergic | 1.1 | 0 | 0.8

2. Secondary Outcome: Event-Free Survival (EFS) as Assessed by Investigator According to International Working Group (IWG) Response Criteria
Description: EFS is defined as the time from first dose of rituximab (analysed using both first dose of IV and first dose of SC) to first occurrence of progression or relapse, according to the IWG response criteria or other country standards, or initiation of a non-protocolspecified anti-lymphoma therapy or death, whichever occurs first.
Time Frame: From first dose of rituximab intravenous (IV) and SC until first occurrence of progression or relapse (up to end of induction treatment [Up to 53.8 Months])
Population: ITT
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Overall: All participants received rituximab SC 1400 milligrams (mg) once a month for a minimum of 4 cycles as induction therapy. Participants with FL will continue to receive rituximab once in 2 months for a minimum of 6 cycles as maintenance therapy according to local standards of care. Participants will also receive standard chemotherapy regimen (CHOP [cyclophosphamide+doxorubicin+vincristine+prednisone], CVP [cyclophosphamide+vincristine+prednisone] or FC [fludarabine+cyclophosphamide]) during induction.
Arm/Group | DLBCL Arm | FL Arm | Overall
Number analyzed (Participants) | 105 | 34 | 139
Months
  From first dose of rituximab IV | NA [33.4 to NA] — The median and upper limit of 95% CI was not evaluable due to an insufficient number of participants with events. | 53.8 [32.6 to NA] — The upper limit of 95% CI was not evaluable due to an insufficient number of participants with events. | 53.8 [38.4 to NA] — The upper limit of 95% CI was not evaluable due to an insufficient number of participants with events.
  From first dose of rituximab SC | NA [32.7 to NA] — The median and upper limit of 95% CI was not evaluable due to an insufficient number of participants with events. | 45.5 [25.1 to NA] — The upper limit of 95% CI was not evaluable due to an insufficient number of participants with events | 45.5 [33.5 to NA] — The upper limit of 95% CI was not evaluable due to an insufficient number of participants with events

3. Secondary Outcome: Progression-Free Survival (PFS) as Assessed by Investigator According to IWG Response Criteria
Description: PFS is defined as the time from first dose of rituximab (analysed using both first dose of IV and first dose of SC) to the first occurrence of progression or relapse, according to the IWG response criteria (Cheson et al. 1999) or other country standards, or death from any cause.
Time Frame: From first dose of rituximab IV and SC until first occurrence of progression or relapse (up to end of induction treatment [Up to 53.8 Months])
Population: ITT
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Overall Population: Participants received rituximab SC 1400 milligrams (mg) once a month for a minimum of 4 cycles as induction therapy. Participants with FL will continue to receive rituximab once in 2 months for a minimum of 6 cycles as maintenance therapy according to local standards of care. Participants will also receive standard chemotherapy regimen (CHOP [cyclophosphamide+doxorubicin+vincristine+prednisone], CVP [cyclophosphamide+vincristine+prednisone] or FC [fludarabine+cyclophosphamide]) during induction
Arm/Group | DLBCL Arm | FL Arm | Overall Population
Number analyzed (Participants) | 95 | 27 | 122
Months
  From first dose of rituximab IV | NA [33.4 to NA] — The median and upper limit of 95% CI was not evaluable due to an insufficient number of participants with events. | 53.8 [32.6 to NA] — The upper limit of 95% CI was not evaluable due to an insufficient number of participants with events. | 53.8 [38.4 to NA] — The upper limit of 95% CI was not evaluable due to an insufficient number of participants with events.
  From first dose of rituximab SC | NA [32.7 to NA] — The median and upper limit of 95% CI was not evaluable due to an insufficient number of participants with events. | 45.5 [25.1 to NA] — The upper limit of 95% CI was not evaluable due to an insufficient number of participants with events. | 44.5 [35.5 to NA] — The upper limit of 95% CI was not evaluable due to an insufficient number of participants with events.

4. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from first dose of rirtuximab (analysed using both first dose of IV and first dose of SC) until death from any cause.
Time Frame: From first dose of rituximab IV and SC until death from any cause (up to end of induction treatment [Up to 51.1 Months])
Population: ITT
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Overall Population: All participants received rituximab SC 1400 milligrams (mg) once a month for a minimum of 4 cycles as induction therapy. Participants with FL will continue to receive rituximab once in 2 months for a minimum of 6 cycles as maintenance therapy according to local standards of care. Participants will also receive standard chemotherapy regimen (CHOP [cyclophosphamide+doxorubicin+vincristine+prednisone], CVP [cyclophosphamide+vincristine+prednisone] or FC [fludarabine+cyclophosphamide]) during induction.
Arm/Group | DLBCL Arm | FL Arm | Overall Population
Number analyzed (Participants) | 95 | 27 | 122
Months
  From first dose of rituximab IV | 51.4 [50.4 to NA] — The upper limit of 95% CI was not evaluable due to an insufficient number of participants with events. | NA [NA to NA] — The median, lower, and upper limit of 95% CI was not evaluable due to an insufficient number of participants with events. | NA [NA to NA] — The median, lower, and upper limit of 95% CI was not evaluable due to an insufficient number of participants with events.
  From first dose of rituximab SC | 51.4 [50.4 to NA] — The upper limit of 95% CI was not evaluable due to an insufficient number of participants with events. | NA [NA to NA] — The median, lower, and upper limit of 95% CI was not evaluable due to an insufficient number of participants with events. | NA [NA to NA] — The median, lower, and upper limit of 95% CI was not evaluable due to an insufficient number of participants with events.

5. Secondary Outcome: Disease-Free Survival (DFS) as Assessed by Investigator According to IWG Response Criteria
Description: DFS will be assessed at the end of induction treatment in patients achieving CR/CRu and is defined as the period from the date of the initial CR/CRu until the date of relapse or death from any cause.
Time Frame: From the date of the initial complete response (CR)/complete response unconfirmed (CRu) until date of relapse or death from any cause (up to end of induction treatment [Up to 32.7 Months])
Population: ITT
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- DLBCL Arm: Participants DLBCL received rituximab SC 1400 milligrams (mg) once a month for a minimum of 4 cycles as induction therapy. Participants with FL will continue to receive rituximab once in 2 months for a minimum of 6 cycles as maintenance therapy according to local standards of care. Participants will also receive standard chemotherapy regimen (CHOP [cyclophosphamide+doxorubicin+vincristine+prednisone], CVP [cyclophosphamide+vincristine+prednisone] or FC [fludarabine+cyclophosphamide]) during induction.
Arm/Group | DLBCL Arm | FL Arm | Overall Population
Number analyzed (Participants) | 95 | 27 | 122
Months | NA [NA to NA] — The median, lower, and upper limit of 95% CI was not evaluable due to an insufficient number of participants with events. | NA [19.7 to NA] — The median and upper limit of 95% CI was not evaluable due to an insufficient number of participants with events. | NA [32.7 to NA] — The median and upper limit of 95% CI was not evaluable due to an insufficient number of participants with events.

6. Secondary Outcome: Percentage of Participants With CR/CRu as Assessed by Investigator According to IWG Response Criteria
Description: CR/CRu: Response assessments 4 - 6 weeks after the last dose of induction treatment will be based on the Investigator's assessment, completed according to the original International Working Group (IWG) response criteria for response assessment of lymphoma (Cheson et al. 1999).
Time Frame: From first dose of rituximab until first occurrence of progression or relapse (up to end of induction treatment [Up to 32 Months])
Population: ITT
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | DLBCL Arm | FL Arm | Overall Population
Number analyzed (Participants) | 95 | 27 | 122
Percentage | 74.2 [63.8 to 82.9] | 76.5 [50.1 to 93.2] | 74.5 [65.1 to 82.5]

7. Secondary Outcome: Healthcare Professional Questionnaire Score
Description: Planned Healthcare Professional Questionnaiere was not collected during the study therefore no data to report
Time Frame: End of treatment (Month 24 for FL participants and Month 8 for DLBCL participants)
Groups:
- Overall Population: Participants with FL and DLBCL will receive rituximab SC 1400 milligrams (mg) once a month for a minimum of 4 cycles as induction therapy. Participants with FL will continue to receive rituximab once in 2 months for a minimum of 6 cycles as maintenance therapy according to local standards of care. Participants will also receive standard chemotherapy regimen (CHOP [cyclophosphamide+doxorubicin+vincristine+prednisone], CVP [cyclophosphamide+vincristine+prednisone] or FC [fludarabine+cyclophosphamide]) during induction.
Arm/Group | Overall Population
Number analyzed (Participants) | 0

8. Secondary Outcome: Patient-Reported Rituximab Administration Questionnaire (RASQ) Score
Description: The RASQ measures the overall participant satisfaction and is a 20-item questionnaire measuring the impact of the treatment administration on 5 domains: Physical Impact, Psychological Impact, Impact on Activities of Daily Living, Convenience, and Satisfaction.
  Each question's answer is chosen from 1 (minimum)-5(maximum score indicating less severity) score range.
  For each domain was scored using the following formula:
  Domain score = [(Sum of completed item (question) responses / Number of completed items) - 1] x 100 / (Maximum possible item response value - Minimum possible item response value)
  The final RASQ domains is calculated using the formula:
  RASQ domain score = (Mean of completed item responses - 1) x 25, scores ranging from 1-100 with higher scores indicative of more positive feelings toward therapy. Lower number representing lower satisfaction and higher is the higher satisfaction by the participants.
Time Frame: Up to 53.8 Months
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Groups:
- Overall Population: Participants with FL and DLBCL received rituximab SC 1400 milligrams (mg) once a month for a minimum of 4 cycles as induction therapy. Participants with FL will continue to receive rituximab once in 2 months for a minimum of 6 cycles as maintenance therapy according to local standards of care. Participants will also receive standard chemotherapy regimen (CHOP [cyclophosphamide+doxorubicin+vincristine+prednisone], CVP [cyclophosphamide+vincristine+prednisone] or FC [fludarabine+cyclophosphamide]) during induction.
Arm/Group | DLBCL Arm | FL Arm | Overall Population
Number analyzed (Participants) | 95 | 27 | 122
Scores on a Scale | 70.5 (20.76) | 69.2 (19.83) | 70.2 (20.48)

ADVERSE EVENTS:
Time Frame: From first dose of rituximab IV and SC until death from any cause (up to end of induction treatment [up to 53.8 Months])
Arm/Group | DLBCL Arm | FL Arm
All-Cause Mortality (participants affected / at risk) | 22/95 | 5/27
Serious Adverse Events (participants affected / at risk) | 11/95 | 8/27
Other Adverse Events (participants affected / at risk) | 58/95 | 12/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DLBCL Arm (N=95) | FL Arm (N=27)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Bone Marrow Failure (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac Failure Acute (Cardiac disorders) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 0 (0) | 1 (1)
Rectal Haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Death (General disorders) | 2 (2) | 1 (1)
Mucosal Inflammation (General disorders) | 2 (4) | 0 (0)
Abscess Limb (Infections and infestations) | 0 (0) | 1 (1)
Candida Infection (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis B Reactivation (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Septic Shock (Infections and infestations) | 0 (0) | 1 (1)
Fibula Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Liver Function Test Abnormal (Investigations) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Generalised Tonic-Clonic Seizure (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Haemorrhagic Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DLBCL Arm (N=95) | FL Arm (N=27)
Neutropenia (Blood and lymphatic system disorders) | 41 (91) | 7 (13)
Anaemia (Blood and lymphatic system disorders) | 13 (24) | 4 (8)
Leukopenia (Blood and lymphatic system disorders) | 10 (13) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 9 (14) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 8 (9) | 0 (0)
Mucosal Inflammation (General disorders) | 10 (12) | 2 (2)
Injection Site Erythema (General disorders) | 5 (5) | 2 (2)
Pyrexia (General disorders) | 5 (5) | 1 (1)
Oral Herpes (Infections and infestations) | 5 (6) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 2 (2)
Paraesthesia (Nervous system disorders) | 14 (15) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2016-02-07): https://cdn.clinicaltrials.gov/large-docs/92/NCT02406092/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-04): https://cdn.clinicaltrials.gov/large-docs/92/NCT02406092/SAP_001.pdf